CLINICAL TRIAL: NCT05092724
Title: Is Fetal Hemoglobin a Key for Improvement of Hypoxia and Saving Last Breath in COVID-19 Patient?. A Pilot Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Essamedin Mamdouh Negm, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #:8046-10-10-2021
Record Dates: First submitted 2021-10-19; First posted 2021-10-25 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: interventions — Blood Transfusion, Intrauterine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard protocol of manaegement (No Intervention)
- fetal blood (Active Comparator)
  Interventions: Procedure: fetal blood transfusion

INTERVENTIONS:
Procedure: fetal blood transfusion — transfusion of fetal blood
  Arms: fetal blood

SUMMARY:
In December 2019, a sudden public health incident (the corona virus disease [COVID-19] epidemic) occurred in Wuhan, China.

Clinical features of those with pneumonia include fever and cough, and in many cases a sudden and accelerating respiratory distress originated from interstitial pneumonia . Many hypotheses have explained hypoxemia in COVID-19 patients, such as hyperimmune reaction to viral infection and cytokine storm that leads to serious lung tissue and alveolar damage or even direct viral insult .

Mortality are as high as 15% in critically ill patients requiring intensive care unit admission and oxygen therapy , suggesting an urgent need to try therapeutic interventions in addition to supportive treatment.

There is more than one type of hemoglobin. In adults, Hb A or Adult hemoglobin which is the main hemoglobin in the blood. But there is another type of hemoglobin called fetal hemoglobin. Fetal hemoglobin (hemoglobin F, Hb F, or α2γ2) is the main oxygen carrier protein in the human fetus. and the levels remain high after birth until the baby is roughly 2-4 months old . Hemoglobin F has a different composition from hemoglobin A and higher affinity to oxygen . At birth, hemoglobin F accounts for 50-95% of the infant's hemoglobin and at around 6 months after birth, hemoglobin A becomes the predominant type.The key feature that allows hemoglobin F to bind more strongly to oxygen is by having γ subunits (instead of β, in Hb A for example). 2,3-BPG interacts much more with hemoglobin A than hemoglobin F .

A hypothesis for the low incidence of the COVID-19 infection in pediatric is the presence of fetal hemoglobin (HbF) .

In a preliminary study about the prevalence of hemoglobinopathies in different countries and the mortality rate of COVID-19, it appears that the mortality is lower in countries with a higher prevalence of hemoglobinopathies .

Mice treated with GBT1118 (a compound that enhances the oxygen affinity of hemoglobin) showed a sustained significant increase in SpO2 over 4 h of hypoxia exposure.

People with haemoglobinopathies like sickle cell anemia or beta-thalassemia attributed with high amount of fetal hemoglobin, become mostly asymptomatic or have mild symptoms .

The volume of umbilical cord blood varies from 50 ml to 140 ml with a mean of 85 ml rich in fetal hemoglobin .

Mesenchymal stem cells (MSCs) have been widely used in the clinical setting, not only for autoimmune diseases but also for infectious diseases , and their safety and effectiveness have been well elucidated . As a noninvasive treatment, hUC-MSC therapy is a very effective and promising method for clinical application and promotion to treat severe COVID-19

the investigators offer a solution by increasing fetal hemoglobin by cord blood containing fetal blood transfusion in the critical patients as a trial to combat the course of the disease and minimize the morbidity especially in sever cases who suffer from desaturation until suppression of the immune dysregulation and avoidance of the impending death.

ELIGIBILITY:
Inclusion Criteria:

* Admitted covid 19 patients to the ICU with the following criteria : :

  * Hypoxia (P/F less than 100)
  * Need for high level of oxygenation or ventilatory support
  * Tachypnea, respiratory distress due to hypoxia
  * >50 percent involvement of the lung parenchyma on chest imaging .

    * Serum IL-6 ≥ 5 x upper normal limit of daily increase of >1 time
    * Ferritin >300 ug/L with doubling within 24 hours
    * Ferritin >600 ug/L at presentation
    * LDH >250 U/L
    * Elevated D-dimer (>1 mg/L)

Exclusion Criteria:

* 1- Patients with hemodynamic instability or multiorgan failure 2- Failure to obtain temporary vascular access under ultrasound guidance or due to bleeding tendency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-02-19 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
• To evaluate the effect of increasing fetal hemoglobin protocol on the outcome in patients with fulminant COVID-19 | for 10 cases for each group ( pilot study ) allover about 5 months
  To show how fetal blood transfusion (cord blood ) improve the outcome of COVID 19 patient ( mortality)

SECONDARY OUTCOMES:
To evaluate the effect of increasing fetal hemoglobin protocol on the morbidity of patients with fulminant COVID-19 | allove 5 months . 10 days for each group .
  To show how fetal blood transfusion (cord blood ) improve the morbidity of COVID 19 patient ( ICU days, M.V days ,oxygenation and perfusion parameters )